CLINICAL TRIAL: NCT05096689
Title: Non-operative Treatment of Pediatric Lateral Humeral Condyle Fractures: a Cohort Study of 50 Patients
Brief Title: Non-operative Treatment of Pediatric Lateral Humeral Condyle Fractures
Acronym: NOTICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Fractures Interest Group, Denmark (Other)
Responsible Party: Principal Investigator, Morten Jon Andersen, Consultant Orthopedic Surgeon, Children's Fractures Interest Group, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-21017621
Record Dates: First submitted 2021-10-12; First posted 2021-10-27 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Fracture Humerus; Physeal Fracture
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Intervention Model Description: Prospective, Cohort, Single center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-operative (Experimental): Non-operative treatment of lateral humeral condyle fractures
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Magnetic Resonance Imaging

SUMMARY:
The diagnosis of LHCF is complicated by radiographic inability to show the full extent of the injury into the chondral (unossified) epiphysis. MRI gives a perfect view of these fractures. The safety and feasibility of non-operative treatment based on MRI findings in children with elbow fractures has not been investigated in a Danish setting. If safe and feasible, the use of MRI could dramatically lower the need for surgery in children with LHCF.

DETAILED DESCRIPTION:
The treatment of LHCF has historically most often been surgical with open reduction and fixation. The diagnosis of LHCF is complicated by radiographic inability to show the full extent of the injury into the unossified chondral epiphysis and therefore physicians often opt for open surgical treatment. MRI; however, gives a perfect view of these fractures. This project investigates the safety and feasibility of non-operative treatment of LHCF based on MRI performed without sedation or anesthesia and seeks to dramatically lower the need for surgery. Objectives are to describe functional outcome, radiological healing, secondary fracture displacement and any complications after two years. The investigators hypothesize that undisplaced and minimally displaced LHCF can be treated non-operatively based on MRI findings with good functional outcomes after two years. A cohort study design is used to follow 50 children with LHCF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute Lateral humeral condyle fracture
* Fracture <5 days old
* Fracture with <5 mm of displacement on plain radiographs
* Parental informed consent obtained

Exclusion Criteria:

* Contraindication(s) to performing an MRI
* Unable to participate in follow-up
* Existing bone pathology
* Previous ipsilateral elbow fracture

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Mayo Elbow Performance Score (MEPS) | 2 years
  MEPS consists of three domains; pain, elbow range of motion (ROM) and stability. The total score ranges from 0-100 with higher scores indicating better function. If the total score ranges between 75 and 100, the result is good (satisfactory); 50-74, fair (acceptable); <50, poor (unsatisfactory).

SECONDARY OUTCOMES:
MRI results | 2 weeks
  Proportion of successful MRIs defined as a completed scan with an image quality that is useful for analysis by the radiologist.
  MRI findings. Song classification based on MRI. Scan length (minutes). Any discomforts for the child during the scan.
Radiographic results | 2 years
  Injury radiographs and subsequent radiographs during FU will be read and described by a senior orthopedic surgeon.
Secondary fracture displacement | 2 years
  Any secondary displacement and amount of radiographic displacement (mm) is recorded.
Pain scale (age <5 years) | 2 years
  To quantify pain in the patient age <5 years, the Face, Legs, Activity, Cry, Consolability Scale (FLACC). To quantify pain behaviors in children who may not be able to verbalize the presence or severity of pain FLACC provides a simple framework. The child is observed for at least 2-5 minutes. Legs and body are observed uncovered. Activity is observed and body is assessed for tenseness and tone.
  Assessment of Behavioural Score: 0 = Relaxed and comfortable. 1-3 = Mild discomfort. 4-6 = Moderate pain. 7-10 = Severe discomfort/pain.
Pain scale (age >4 years) | 2 years
  To quantify pain in the patient >4 years, Faces Pain Scale - Revised (FPS-R) is applied.
  The Faces Pain Scale - Revised (FPS-R) is used to quantify pain in children above four years of age. It is a self-report measure of pain intensity developed for children. It was adapted from the Faces Pain Scale to make it possible to score the sensation of pain on a 0-to-10 metric. The scale shows a close linear relationship with visual analog pain scales (VAS) across the age range of 4-16 years.
  FPS-R is easy to administer and requires no equipment except for the photocopied faces. The child is asked to point to the face that shows how much pain the child is in at that moment. Faces are scored 0-10 so 0 equals no pain and 10 equals very much pain.
Pain scale (age >8 years) | 2 years
  A visual analogue scale (VAS) is used to quantify pain in children age 8 and above. VAS has been extensively investigated in quantifying pain in older children. The child is asked to put a mark on the line corresponding to the child's pain at that moment. A mark to the far left equals no pain and a mark to the far right equals worst possible pain. The line is 10 cm long and the child's mark is measured from left to right in cm with one decimal e.g., 3.4 cm equaling a VAS of 3.4. If the child cannot cooperate to using VAS, FPS-R is used instead.

CONTACTS AND LOCATIONS:
Overall Officials: Morten J Andersen, MD, Principal Investigator
Locations (1):
- Copenhagen University Hospital - Herlev and Gentofte, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT05096689/Prot_000.pdf